CLINICAL TRIAL: NCT05389098
Title: L'Alimentation Manger-mains, le Plaisir au Bout Des Doigts : Etude Pilote randomisée, en Ouvert et en Groupes parallèles
Brief Title: Finger Food, Pleasure at Your Fingertips: Randomized Pilot Study, Open-label and Parallel Groups
Acronym: PLAID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DR200176-PLAID; ID-RCB (Registry Identifier: 2021-A01094-37)
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Undernutrition; Elderly Person
Keywords: Undernutrition; Elderly Person; Nursing home; Nutrition
MeSH Terms: conditions — Malnutrition | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Pilot Study, Open-label and Parallel Groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): eat-hands type food mode
  Interventions: Other: Hand-Eating
- Control (Active Comparator): Usual food administration
  Interventions: Other: Control

INTERVENTIONS:
Other: Hand-Eating — eat-hands type food mode
  Other Names: EXPERIMENTAL
  Arms: Experimental
Other: Control — Usual eating mode
  Other Names: Control group
  Arms: Control

SUMMARY:
Food is available in easy-to-grip bites that allow residents in care settings to use their fingers for food. This new way of eating can help limit weight loss, increase food intake, gain independence and improve the enjoyment of eating for residents.

DETAILED DESCRIPTION:
According to the Haute Autorité de Santé (HAS), undernutrition affects between 15 and 38% of elderly people living in institutions and between 50 and 60% of hospitalized elderly people. In addition, a significant decrease in satisfaction with meals was observed with increasing level of dependence.

The objective of the study is to evaluate the feasibility of implementing the finger food in care settings that could have a positive impact on the nutritional status of elderly people living in EHPAD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female residents over 75 years old living in a Accommodation facility for dependent elderly people for at least 3 months
* Presenting at least one of the following 3 criteria:

  * Unintentional weight loss ≥ 5% in 1 month
  * Involuntary weight loss ≥ 10% in 6 months or compared to the usual weight or compared to the weight at entry to the EHPAD
  * Confirmed sarcopenia:

    * Male (at least one of the 2 criteria):

      * Dynamometer (kg): < 27 AND calf circumference (cm): < 31
      * Impedancemetry: appendicular muscle mass index < 20 kg OR appendicular muscle mass index < 7 kg/m²
    * Woman (at least one of the 2 criteria):

      * Dynamometer (kg): < 16 AND calf circumference (cm): < 31
      * Impedancemetry: appendicular muscle mass index < 15 kg OR appendicular muscle mass index < 5.5 kg/m²
* Loss of autonomy according to the Tully scale < 12/18 with a score of 2 or 3 on the item "Able to bite, chew, swallow without making false routes"
* Person having given free, informed and express consent
* Person having an affiliation to a social security scheme

Exclusion Criteria:

* Protected person: safeguard of justice
* Swallowing disorder having a contra-indication to the texture of hand-eating meals.
* Lack of motor skills in both hands
* Specific diet: pleasure diet, salt-free, sugar-free, fiber-free, artificial nutrition
* Wearer of a pacemaker

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Audit & Questionnaire of feasibility | After 3 patients included and at the end of study (6 months)
  Feasibility of implementing finger food for elderly patients in care settings will be evaluate with audit and questionnaire for caregivers by a dietician independent of the study.

SECONDARY OUTCOMES:
Weight | Every two weeks during 6 months
  Weight in kilograms
Food consumption | Each week during 6 months
  Each week, a semi-quantitative evaluation of food intake will be performed for 3 days on a specific form (validated by the Francophone Society of Clinical and Metabolic Nutrition ). Every month, dietician will analyze these forms.
Autonomy (EBS) | Every month during 6 months
  Autonomy for food intake will be assessed by the Eating Behavior Scale - EBS (Tully MW, Matrakas KL, Muir J, Musallam K. The Eating Behavior Scale. A simple method of assessing functional ability in patients with Alzheimer's disease. J Gerontol Nurs. 1997 Jul;23(7):9-15; quiz 54-5. doi: 10.3928/0098-9134-19970701-08. PMID: 9287601) by a dietetician.
  The scores on this scale range from 0 to 18 : 18 is the best score, which means that the person is completely independent in eating.
Eating pleasure | Every month during 6 months
  An evaluation of the pleasure of eating will be carried out once a month by the dietician via an hedonic scale with 3 face symbols: smiling face - neutral face - disappointed face.
False routes | Every week during 6 months
  The occurrence of false routes will be collected throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Laura COUTON, Study Director — CHU Tours; Laura COUTON, Principal Investigator — CHU Tours
Locations (2):
- France (2):
  - EHPAD " Val de Brenne " Site : Auzouer en Touraine, Château-Renault
  - EHPAD L'ERMITAGE-CHU de TOURS, Tours

IPD SHARING:
Plan to Share IPD: No